CLINICAL TRIAL: NCT05881317
Title: Intra-Articular Hyaluronic Acid (ArtiAid® Plus) for Knee Osteoarthritis: A Post-market, Open-Label, Long-Term Historical Control Study
Brief Title: ArtiAid® Plus for Knee Osteoarthritis: A Post-market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MCQ-200305
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hyaluronic Acid
Keywords: Viscosupplements; Osteoarthritis, Knee; Injections, Intra-Articular
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ArtiAid® Plus group (Experimental): Each pre-filled syringe contains 15 mg/ml (1.5%) sodium hyaluronate, subjects received one injection per week for three weeks.
  Interventions: Device: ArtiAid® Plus Intra-articular Injection

INTERVENTIONS:
Device: ArtiAid® Plus Intra-articular Injection — Inject ArtiAid® Plus in the affected joint at weekly interval for 3 weeks

SUMMARY:
The goal of this open-label, post-market clinical follow-up study is to demonstrate the safety and performance of ArtiAid® Plus Intra-articular Injection in patients with knee osteoarthritis(OA). The main questions it aims to answer are:

* the safety profile of ArtiAid® Plus;
* the clinical performance of ArtiAid® Plus, such as pain relief and satisfaction of treatment.

Participants will receive weekly injections of ArtiAid® Plus for 3 weeks and be follow-up for 26 weeks.

DETAILED DESCRIPTION:
An open-label study will be performed in single center to monitor about 60 patients with knee osteoarthritis(OA), each treated with 3 injections of ArtiAid® Plus 1.5% (MAXIGEN BIOTECH INC., Taiwan). Follow-up visits will be at 4 weeks, 12 weeks(a telephone contact by the investigator) and 26 weeks after the injections. The primary endpoint of this study is to monitor the adverse events after injecting ArtiAid® Plus. The secondary endpoints of this study are demonstrating the clinical performance of ArtiAid® Plus, such as resting knee pain and satisfaction of treatment by using the visual analog scale (VAS). Analysis of variance (ANOVA) will be applied to the clinical data and T-test will be used to test for the differences between baseline and each visit. The paired student t-test was used to analyze variations in each group over a period of time. Statistical significance was established at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged older than 40 years old.
* Able to sign informed consent prior to the study.
* Subjects have Kellgren-Lawrence (KL) grade 2 to 3 knee osteoarthritis.
* Subjects have failed to respond adequately to conservative non-pharmacological therapy.
* Plasma pregnancy test at screening visit must be negative for fertile female subjects.
* Subjects in stable progress of disease as judged by the investigator.

Exclusion Criteria:

* Subjects with known hypersensitivity to hyaluronate preparations.
* Subjects with infections or skin diseases in the area of the injection site.
* Pregnancy or breast-feeding woman.
* Significant drug, alcohol abuse.
* Joining any clinical trial within 3 months prior to dosing.
* Subjects have traveled abroad within 3 months prior to the screening visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 0 week to 26 weeks after injections
  The adverse events are defined as any unfavorable sign occurrence in a subject after treatment. The investigator assesses the severity and the relationship of each event to the use of the study device.

SECONDARY OUTCOMES:
Resting knee pain: VAS (visual analog scale) | Baseline, 4 weeks, and 26 weeks after injections
  Current level of resting knee pain will be assessed by a patient-reported VAS (visual analog scale), subjects mark on a 0-100 mm line, where 0 represent "no pain" and 100 represents "maximum pain". The VAS pain score will be assessed at baseline 4 weeks and 26 weeks after injections.
Satisfaction of treatment: VAS (visual analog scale) | 4 weeks, and 26 weeks after injections
  The satisfaction of treatment will be assessed by a patient-reported VAS (visual analog scale), subjects mark on a 0-100 mm line, where 0 represent "least satisfied" and 100 represents "highest satisfaction". The VAS pain score will be assessed at 4 weeks and 26 weeks after injections.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Fong Chen, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Maxigen Biotech Inc., Taoyuan, Taiwan (r.o.c.), Taiwan

REFERENCES:
- [Derived] Chen CF, Chen CT, Lin YH, Chiang CF, Mao YW. Safety and clinical performance of intra-articular high-purity sodium hyaluronate injection in patients with knee osteoarthritis: a 28-week post-market clinical follow-up study. Clin Rheumatol. 2025 Dec 24. doi: 10.1007/s10067-025-07891-1. Online ahead of print. PMID 41436701